CLINICAL TRIAL: NCT06213818
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Single-Dose, Dose-Escalation, Drug-Interaction, and Food-Effect Study to Assess the Safety, Tolerability, and Pharmacokinetics of INCB160058 When Administered Orally to Healthy Adult Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of INCB160058 When Administered Orally to Healthy Adult Participant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB160058-102
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants
Keywords: INCB160058
MeSH Terms: interventions — Esomeprazole; Famotidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- Cohort 1: Dose (Experimental): INCB160058 or placebo will be administered at protocol defined dose after an overnight fast.
  Interventions: Drug: INCB160058; Drug: Placebo
- Cohort 2: Dose (Experimental): INCB160058 or placebo will be administered at protocol defined dose after an overnight fast.
  Interventions: Drug: INCB160058; Drug: Placebo
- Cohort 3: Dose (Experimental): INCB160058 or placebo will be administered at protocol defined dose after an overnight fast.
  Interventions: Drug: INCB160058; Drug: Placebo
- Cohort 4: Dose (Experimental): INCB160058 or placebo will be administered at protocol defined dose after an overnight fast.
  Interventions: Drug: INCB160058; Drug: Placebo
- Cohort 5: Dose (Experimental): INCB160058 or placebo will be administered at protocol defined dose after an overnight fast.
  Interventions: Drug: INCB160058; Drug: Placebo
- Cohort 6: Dose Treatment A (Experimental): INCB160058 will be administered at protocol defined dose after an overnight fast.
  Interventions: Drug: INCB160058
- Cohort 6: Dose Treatment B (Experimental): INCB160058 will be administered at protocol defined dose after a high-fat, high-calorie meal.
  Interventions: Drug: INCB160058
- Cohort 7: Dose (Experimental): INCB160058 and esomeprazole will be administered at protocol defined schedule and dose.
  Interventions: Drug: INCB160058; Drug: Esomeprazole
- Cohort 8: Dose (Experimental): INCB160058 will be administered at protocol defined dose after an overnight fast.
  Interventions: Drug: INCB160058
- Cohort 9: Dose (Experimental): INCB160058 or placebo will be administered at protocol defined dose after an overnight fast.
  Interventions: Drug: INCB160058; Drug: Placebo
- Cohort 10: Dose Treatment A (Experimental): INCB160058 will be administered at protocol defined dose after an overnight fast.
  Interventions: Drug: INCB160058
- Cohort 10: Dose Treatment B (Experimental): INCB160058 will be administered at protocol defined dose after a high-fat, high-calorie meal.
  Interventions: Drug: INCB160058
- Cohort 11: Dose (Experimental): INCB160058 and esomeprazole will be administered at protocol defined schedule and dose.
  Interventions: Drug: INCB160058; Drug: Esomeprazole
- Cohort 12: Dose (Experimental): INCB160058 and famotidine will be administered at protocol defined schedule and dose.
  Interventions: Drug: INCB160058; Drug: Famotidine
- Cohort 13: Dose (Experimental): INCB160058 or placebo will be administered at protocol defined dose after an overnight fast.
  Interventions: Drug: INCB160058; Drug: Placebo
- Cohort 14: Dose (Experimental): INCB160058 and famotidine will be administered at protocol defined schedule and dose.
  Interventions: Drug: INCB160058; Drug: Famotidine
- Cohort 15: Dose (Experimental): INCB160058 or placebo will be administered at protocol defined dose after an overnight fast.
  Interventions: Drug: INCB160058; Drug: Placebo

INTERVENTIONS:
Drug: INCB160058 — Oral; Immediate release solid tablet
Drug: Placebo — Oral; Tablet
  Arms: Cohort 13: Dose; Cohort 15: Dose; Cohort 1: Dose; Cohort 2: Dose; Cohort 3: Dose; Cohort 4: Dose; Cohort 5: Dose; Cohort 9: Dose
Drug: Esomeprazole — Oral; Delayed-release capsule or tablet
  Arms: Cohort 11: Dose; Cohort 7: Dose
Drug: Famotidine — Oral; Tablet
  Arms: Cohort 12: Dose; Cohort 14: Dose

SUMMARY:
This study is being conducted to assess the Safety, Tolerability, and Pharmacokinetics of INCB160058 When Administered Orally to Healthy Adult Participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Age 18 to 55 years, inclusive, at the time of signing the ICF.
* Body mass index between 18.0 and 32.0 kg/m2 (inclusive).
* Willingness to adhere to study-related prohibitions, restrictions, and procedures.
* Ability to swallow and retain oral medication.
* Willingness to avoid pregnancy or fathering children based on the criteria below.

  * Male participants with reproductive potential must agree to use 1 of the highly effective methods of contraception to avoid fathering children from screening through the last follow-up visit and must refrain from donating sperm during this period. Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Female participants who are WOCBP must have a negative pregnancy test at screening and check-in, must agree to use 1 of the highly effective methods of contraception to avoid pregnancy from screening through the last follow-up visit, and must refrain from donating oocytes during this period.

Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed. Positive pregnancy tests may be confirmed at the investigator's discretion.

• Female participants not considered to be of childbearing potential are eligible and must have a negative pregnancy test at screening and check-in.

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening.
* History of rheumatologic/autoimmune disorders and immune deficiency/immunologic defects.
* Prior history of major bleeding or thrombosis, including myocardial infarction/stroke and pulmonary embolism/deep vein thrombosis.
* Known tuberculosis infection that is active or participant-reported history of tuberculosis or treatment thereof.
* Resting pulse < 40 bpm or > 100 bpm, confirmed by repeat testing at screening.
* History or presence of an abnormal ECG before initial dose administration that, in the investigator's opinion, is clinically significant (QTcF interval > 450 milliseconds, QRS interval > 120 milliseconds, and PR interval > 220 milliseconds).
* Presence of a malabsorption syndrome possibly affecting drug absorption (eg, Crohn disease or chronic pancreatitis).
* Hemoglobin level, WBC count, platelet count, or absolute neutrophil count below the laboratory lower limit of normal at screening or at check-in, confirmed by repeat testing and clinically significant in the opinion of the investigator.
* Hepatic transaminase (ALT and AST), ALP, or total bilirubin levels > 1.25 × the laboratory-defined ULN at screening or at check-in, confirmed by repeat testing (except participants with Gilbert disease, for which total bilirubin must be ≤ 2.0 × ULN).
* History of malignancy within 5 years of screening, with the exception of cured basal cell or squamous cell carcinoma of the skin, ductal carcinoma in situ, or prostate cancer.
* Current or recent (within 3 months of screening) clinically significant gastrointestinal disease or surgery (including cholecystectomy) that could affect the absorption of study drug, with the exception of appendectomy.
* Any major surgery within 12 weeks of screening.
* Donation of blood to a blood bank within 4 weeks of screening (within 2 weeks for plasma only).
* Blood transfusion within 4 weeks of check-in.
* Chronic or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment.
* Positive test for hepatitis B virus, hepatitis C virus, or human immunodeficiency virus.

Note: Participants whose results are compatible with prior immunization or immunity due to infection for hepatitis B may be included at the discretion of the investigator.

* Regular alcohol consumption > 21 units per week (1 unit = ½ pint beer or a 25-mL shot of 40% spirit, 1.5 to 2 units = 125-mL glass of wine, depending on type).
* Positive urine or breath test for ethanol or positive urine or serum screen for drugs of abuse that are not otherwise explained by permitted concomitant medications or diet.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with another investigational medication or current enrollment in another investigational drug protocol.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with an inducer or inhibitor of CYP3A4, P-gp, or BCRP (refer to the Drug Interaction Database for prohibited drugs).
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) deemed clinically relevant by the investigator.
* Known hypersensitivity or severe reaction to INCB160058 or any excipients of INCB160058 (refer to the IB).
* Inability to undergo venipuncture or tolerate venous access.
* Inability or unlikeliness of the participant to comply with the dose schedule and study evaluations, in the opinion of the investigator.
* Use of tobacco- or nicotine-containing products within 1 month of screening.
* Use of prescription drugs (including oral, implantable, transdermal, injectable, intravaginal, or hormonal intrauterine contraceptives) or topical steroids within 14 days prior to study drug administration or nonprescription medications/products (including vitamins, minerals, and phytotherapeutic, herbal, or plant-derived preparations) within 7 days prior to study drug administration and during the study.

Note: Occasional use of acetaminophen (see Section 6.6.1) is permitted during the study.

* Women who are pregnant or breastfeeding.
* eGFR < 90 mL/min/1.73 m2 based on the Chronic Kidney Disease Epidemiology Collaboration formula.
* Any history of hypersensitivity or intolerance to esomeprazole or any other PPI, or to famotidine or any other H2 antagonist.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study treatment and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) | Up to Day 28
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
INCB160058 pharmacokinetic (PK) when administered as solid tablets in Plasma | Up to Day 5
  INCB160058 concentration in plasma.
INCB160058 pharmacokinetic (PK) when administered as a soft gel capsule in Plasma | Up to Day 5
  INCB160058 concentration in plasma.
INCB160058 pharmacokinetic (PK) when administered as ASD tablets in Plasma | Up to Day 5
  INCB160058 concentration in plasma.
INCB160058 pharmacokinetic (PK) in Plasma to determine the effect of food administered as solid tablets | Up to Day 12
  INCB160058 concentration in plasma.
INCB160058 pharmacokinetic (PK) in Plasma to determine the effect of food administered as ASD tablets | Up to Day 12
  INCB160058 concentration in plasma.
INCB160058 pharmacokinetic (PK) in Plasma to assess the effect of esomeprazole administered as solid tablets | Up to Day 14
  INCB160058 concentration in plasma.
INCB160058 pharmacokinetic (PK) in Plasma to assess the effect of esomeprazole administered as ASD tablets | Up to Day 14
  INCB160058 concentration in plasma.
INCB160058 pharmacokinetic (PK) in Plasma to assess the effect of famotidine administered as solid tablets | Up to Day 14
  INCB160058 concentration in plasma.
INCB160058 pharmacokinetic (PK) in Plasma to assess the effect of famotidine administered as ASD tablets | Up to Day 14
  INCB160058 concentration in plasma.

SECONDARY OUTCOMES:
Additional INCB160058 pharmacokinetic (PK) in Plasma | Up to Day 14
  Additional INCB160058 concentration in plasma.
INCB160058 pharmacokinetic (PK) in Urine | Up to Day 5
  INCB160058 concentration in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical, Study Director — Incyte Corporation
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of INCB160058 When Administered Orally to Healthy Adult Participant — https://www.incyteclinicaltrials.com/study/?id=INCB160058-102&SearchTerm=INCB160058-102&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=